CLINICAL TRIAL: NCT04027803
Title: A Double-blind, Randomized Clinical Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of Single Intravenous Doses of BCD-148 (JSC BIOCAD, Russia) and Soliris® in Healthy Volunteers
Brief Title: Comparative Study of Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of Single Intravenous Doses of BCD-148 and Soliris®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-148-3
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-148 (Experimental): 39 healthy subjects received BCD-148, 900 mg, a single drip infusion over 25-45 min
  Interventions: Biological: BCD-148
- Soliris (Active Comparator): 39 healthy subjects received Soliris, 900 mg, a single drip infusion over 25-45 min
  Interventions: Biological: Soliris

INTERVENTIONS:
Biological: BCD-148 — single intravenous infusion of BCD-148 (900 mg)
  Other Names: eculizumab
  Arms: BCD-148
Biological: Soliris — single intravenous infusion of Soliris (900 mg)
  Other Names: eculizumab
  Arms: Soliris

SUMMARY:
A Double-blind, Randomized Clinical Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety, and Immunogenicity of Single Intravenous Doses of BCD-148 (JSC BIOCAD, Russia) and Soliris® in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF for participation in the study
2. Men from 18 to 45 years old (inclusive) at the time of signing the ICF
3. BMI within the normal limits (18.0 to 30 kg/m2)
4. The subject is able to follow the Protocol procedures (in the investigator's opinion)
5. The subject is verified as "Healthy" according to results of standard clinical, laboratory and instrumental tests
6. Normal hemodynamic parameters: systolic BP from 90 mmHg to 130 mmHg; diastolic BP from 60 mmHg to 90 mmHg; HR from 60 bpm to 90 bpm
7. The subject and his sex partner of childbearing potential consent to implement reliable contraceptive methods from the moment the subject signs the ICF and until the subject completes the study. This requirement does not apply to those subjects who had undergone surgical sterilization. Reliable contraception methods mean one barrier method in combination with one of the following: spermicides, intrauterine device and/or oral contraceptives used by the subject's partner.
8. The subject agrees not to drink alcohol for 24 h prior to the infusion of the test/reference drug and for the entire period while the subject is in the study.

   -

Exclusion Criteria:

1. Psychiatric disorders or other conditions that can affect the ability of the subject to follow the study protocol
2. Acute infections within 4 weeks before signing the ICF
3. Results of laboratory and/or instrumental tests are outside the site's normal range
4. Any surgery done within 30 days before the screening or planned within 30 days after the subject completes the study
5. Impossibility to insert an intravenous catheter for blood collection (e.g., because of a skin condition at the venipuncture site)
6. A history of allergies
7. Known hypersensitivity to any component of BCD-148 or Soliris®, murine proteins or other drug components; hypersensitivity to any component of the meningococcal vaccine
8. The subject had used any medications that significantly affect hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) within 30 days before signing the ICF and/or the subject needs any medications (other than the study drugs) to be taken during the entire study period
9. The subject had previously used eculizumab and/or other therapeutic monoclonal antibodies against complement C5
10. Regular use (oral or parenteral) of any drugs, including OTC products, vitamins or biologically active supplements within 14 calendar days before signing the ICF
11. A history of recurrent/chronic hemorrhages or any hemorrhage within 30 days prior to signing the ICF
12. Acute or chronic infections or other diseases that, in the investigator's opinion, may affect the PK, PD or safety of the study products
13. HIV, HCV, HBV infection, syphilis.
14. Meningococcal infection in the past (documented or mentioned verbally by the subject)
15. Vaccination within 4 weeks before the planned infusion date, except for vaccination against Neisseria meningitidis given to all subjects in the screening period
16. The subject refuses to get a vaccination against Neisseria meningitidis during the screening period .
17. The subject smokes more than 10 cigarettes per day
18. The subject consumes more than 10 units of alcohol per week (1 unit equals to 0.5 L of beer, 200 mL of wine or 50 mL of a strong alcohol beverage) or has a history of alcohol, recreational drug or medication abuse, or tests positive for alcohol and/or psychoactive substances during the screening examination
19. Donation of ≥ 450 mL of blood or plasma within 60 calendar days before signing the ICF.
20. Participation in any drug clinical studies within 30 calendar days prior to signing the informed consent form and through the entire period of study participation.

    -

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2019-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company Research Center Eco-Bezopasnost (OOO Research Center Eco-Bezopasnost), Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-148: 39 healthy subjects/ BCD-148: single 900 mg drip infusion given over 25-45 min
  BCD-148: single intravenous infusion of 900 mg BCD-148 active substance of BCD-148 is eculizumab - a monoclonal antibody that targets complement protein C5
- Soliris: 39 healthy subjects Soliris: single 900 mg drip infusion given over 25-45 min
  Soliris: single intravenous infusion of 900 mg BCD-148 active substance of Soliris is eculizumab - a monoclonal antibody that targets complement protein C5
Period: Overall Study
Arm/Group | BCD-148 | Soliris
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BCD-148: 39 healthy subjects BCD-148: single 900 mg drip infusion given over 25-45 min
  BCD-148: single intravenous infusion of 900 mg BCD-148 active substance of BCD-148 is eculizumab - a monoclonal antibody that targets complement protein C5
- Total: Total of all reporting groups
Arm/Group | BCD-148 | Soliris | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [24 to 32] | 27 [24 to 32] | 27 [24 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 39 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 39 | 39 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞ of Eculizumab
Description: AUC0-∞ of eculizumab (the area under the Concentration vs. Time curve from 0 to infinity)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
(ng/ml)*hour | 104346442.41 [86711718.872 to 138234664.3] | 114291981.79 [95801210.959 to 126281914.98]

2. Secondary Outcome: Cmax of Eculizumab
Description: Cmax of eculizumab (maximum concentration of eculizumab in the serum)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
ng/ml | 102466648.13 [86216316.914 to 130773188.67] | 112710712.24 [95318606.352 to 125562084.16]

3. Secondary Outcome: Тmax of Eculizumab
Description: Тmax of eculizumab (time to Cmax)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
hour | 8 [4 to 12] | 8 [0.083 to 24]

4. Secondary Outcome: AUC0-1392 of Eculizumab
Description: AUC0-1392 of eculizumab (the area under the Concentration vs. Time curve from 0 to 1392 h post-infusion)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
(ng/ml)*hour | 102466648.13 [86216316.914 to 130773188.67] | 112710712.24 [95318606.352 to 125562084.16]

5. Secondary Outcome: Т1/2 of Eculizumab
Description: Т1/2 of eculizumab (half-life)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
hour | 165.429 [154.479 to 198.042] | 161.61 [132.711 to 209.22]

6. Secondary Outcome: Vd of Eculizumab
Description: Vd of eculizumab (steady-state volume of distribution)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
ml | 2595.302 [2118.734 to 3434.689] | 2620.503 [1973.187 to 2984.036]

7. Secondary Outcome: Кel of Eculizumab
Description: Кel of eculizumab (elimination constant)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: 1/h
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
1/h | 0.004 [0.004 to 0.004] | 0.004 [0.003 to 0.005]

8. Secondary Outcome: Cl of Eculizumab
Description: Cl of eculizumab (clearance)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: ml/(h*kg)
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
ml/(h*kg) | 8.783 [6.882 to 10.439] | 7.985 [7.168 to 9.442]

9. Secondary Outcome: ABEC(0-1392) CH50
Description: ABEC(0-1392) CH50 (the area between the baseline and effect curves for hemolytic activity of serum complement from 0 to 1392 h)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: (%)*h
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
(%)*h | -33606.865 [-51185.201 to -20772.736] | -37244.026 [-49459.807 to -25247.772]

10. Secondary Outcome: AUEC(0-1392) CH50
Description: AUEC(0-1392) CH50 ((area under the Time vs. Effect curve from 0 to 1392 h)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: (%)*h
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
(%)*h | 61600.835 [45529.369 to 75529.787] | 53479.141 [40111.132 to 72474.492]

11. Secondary Outcome: Emin CH50
Description: Emin CH50 (minimum hemolytic complement activity from 0 to 1392 h)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: % of hemolitic activity
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
% of hemolitic activity | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: Tmin CH50
Description: Tmin CH50 (time to minimum hemolytic complement activity within the period from 0 to 1392 h)
Time Frame: from 0 to 1392 hours post-infusion
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
hour | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.083]

13. Secondary Outcome: Subjects With AEs/SAEs Related to Eculizumab
Description: The percentage of subjects with AEs/SAEs that, in the investigator's opinion, are related to eculizumab
Time Frame: from 0 to 1392 hours post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
Participants | 28 | 30

14. Secondary Outcome: Subjects Who Develop Grade 3/4 AEs Related to Eculizumab
Description: • The percentage of subjects with СТСАЕ v. 4.03 grade 3/4 AEs that, in the investigator's opinion, are related to eculizumab, by study arms.
Time Frame: from 0 to 1392 hours post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-148 | Soliris
Number analyzed (Participants) | 39 | 39
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: 82 days
Arm/Group | BCD-148 | Soliris
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 28/39 | 31/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-148 (N=39) | Soliris (N=39)
anemia (Blood and lymphatic system disorders) | 7 | 9
eosinophils count increase (Blood and lymphatic system disorders) | 2 | 1
lymphocytosis (Blood and lymphatic system disorders) | 5 | 4
lymphopenia (Blood and lymphatic system disorders) | 4 | 6
monocytes count increase (Blood and lymphatic system disorders) | 3 | 0
neutropenia (Blood and lymphatic system disorders) | 11 | 9
platelet count decrease (Blood and lymphatic system disorders) | 1 | 2
ESR increase (Investigations) | 14 | 10
INR decrease (Investigations) | 5 | 7
prothrombin time decreased (Investigations) | 5 | 7
prothrombin time increased (Investigations) | 2 | 1
leukopenia (Blood and lymphatic system disorders) | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04027803/Prot_SAP_001.pdf